CLINICAL TRIAL: NCT00438958
Title: A Randomized Multicentre Study Comparing G-CSF Mobilized Peripheral Blood and G-CSF Stimulated Bone Marrow in Patients Undergoing Matched Sibling Transplantation for Hematologic Malignancies
Brief Title: Sibling Donor Peripheral Stem Cell Transplant or Sibling Donor Bone Marrow Transplant in Treating Patients With Hematologic Cancers or Other Diseases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Canadian Blood and Marrow Transplant Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000528289; CBMTG-0601
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Leukemia; Lymphoma; Myelodysplastic Syndromes; Secondary Myelofibrosis
Keywords: graft versus host disease; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; refractory anemia with ringed sideroblasts; refractory anemia; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; refractory chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; primary myelofibrosis; secondary myelofibrosis; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent small lymphocytic lymphoma; splenic marginal zone lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; Waldenström macroglobulinemia; secondary acute myeloid leukemia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Leukemia; Lymphoma; Myelodysplastic Syndromes; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory; Leukemia, Myelomonocytic, Chronic; Leukemia, Lymphocytic, Chronic, B-Cell; Primary Myelofibrosis; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Waldenstrom Macroglobulinemia | interventions — Filgrastim; Peripheral Blood Stem Cell Transplantation

ARMS (2):
- Arm I (Active Comparator): Patients undergo filgrastim (G-CSF)-mobilized sibling donor peripheral blood SCT on day 0.
  Interventions: Biological: filgrastim; Procedure: peripheral blood stem cell transplantation
- Arm II (Experimental): Patients undergo G-CSF-mobilized sibling donor bone marrow transplantation on day 0.
  Interventions: Biological: filgrastim; Procedure: allogeneic bone marrow transplantation

INTERVENTIONS:
Biological: filgrastim — Given on day 0.
Procedure: allogeneic bone marrow transplantation — Given on day 0
  Arms: Arm II
Procedure: peripheral blood stem cell transplantation — Given on day 0
  Arms: Arm I

SUMMARY:
RATIONALE: Giving chemotherapy before a donor peripheral stem cell transplant or bone marrow transplant using stem cells from a brother or sister that closely match the patient's stem cells, helps stop the growth of cancer or abnormal cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer or abnormal cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving colony-stimulating factors, such as G-CSF, to the donor helps the stem cells move from the bone marrow to the blood so they can be collected and stored. Giving methotrexate and cyclosporine before and after transplant may stop this from happening. It is not yet known whether a donor peripheral stem cell transplant is more effective than a donor bone marrow transplant in treating hematologic cancers or other diseases.

PURPOSE: This randomized phase III trial is studying filgrastim-mobilized sibling donor peripheral stem cell transplant to see how well it works compared with sibling donor bone marrow transplant in treating patients with hematologic cancers or other diseases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the time to treatment failure in patients with hematologic malignancies or other diseases treated with filgrastim (G-CSF)-mobilized matched-sibling donor peripheral blood stem cell transplantation vs G-CSF-stimulated matched-sibling donor bone marrow transplantation.

Secondary

* Compare the hematological recovery and overall survival of patients treated with these regimens.
* Compare the quality of life, in terms of extensive graft-versus-host disease (GVHD), in patients treated with these regimens.
* Compare the economic impact associated with these treatment regimens.

Tertiary

* Compare the incidence and severity of acute GVHD in patients treated with these regimens.
* Compare organ involvement, symptomatology, and functional impact of chronic GVHD in patients treated with these regimens.
* Compare disease-free survival of patients treated with these regimens.
* Compare donor quality of life.
* Compare cost analysis, from a societal perspective, of these treatment regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to treatment center, disease (chronic myelogenous leukemia vs acute myeloid leukemia vs myelodysplastic syndromes vs other hematologic malignancy), disease stage (early disease vs late disease), and conditioning regimen (busulfan and cyclophosphamide vs cyclophosphamide and total body irradiation vs other).

* Myeloablative conditioning regimen: Patients receive a myeloablative conditioning regimen that has been approved by the clinical chair.
* Stem cell transplantation (SCT): Patients are randomized to 1 of 2 SCT arms.

  * Arm I: Patients undergo sibling donor filgrastim (G-CSF)-mobilized peripheral blood SCT on day 0.
  * Arm II: Patients undergo sibling donor G-CSF- mobilized bone marrow transplantation on day 0.
* Graft-verus-host disease (GVHD) treatment: Patients receive methotrexate IV on days 1, 3, 6, and 11 and cyclosporine IV (or orally) every 12 hours beginning on day -2 and continuing until day 100.

Quality of life is assessed at baseline and at 1 and 3 years post-transplantation.

After completion of study therapy, patients are followed periodically for at least 4 years.

PROJECTED ACCRUAL: A total of 230 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following hematologic malignancies:

  * Acute myeloid leukemia in first complete remission or second complete remission
  * Chronic myeloid leukemia in chronic or accelerated phase
  * Myelodysplasia, including any of the following:

    * Refractory anemia (RA)
    * RA with ringed sideroblasts
    * RA with excess blasts (RAEB) I
    * RAEB in transformation
    * Chronic myelomonocytic leukemia
  * Other hematologic malignancy for which sibling donor stem cell transplantation with a myeloablative conditioning regimen is appropriate, including any of the following:

    * Indolent non-Hodgkin's lymphoma (NHL)
    * Aggressive NHL
    * Chronic lymphocytic leukemia
    * Hodgkin's lymphoma
    * Myelofibrosis
    * Hematologic malignancy not otherwise specified
* HLA-matched sibling donor available meeting all of the following criteria:

  * 6/6 HLA match

    * HLA typing performed by serologic or DNA methodology for A and B and by DNA methodology for DRB1 (intermediate resolution)
  * Not identical twin with patient

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No cognitive, linguistic, or emotional difficulty that would preclude participation in the quality-of-life component of the study
* Able to communicate in English or French
* No HIV antibody positivity

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2007-03

PRIMARY OUTCOMES:
Time to treatment failure (extensive chronic graft-versus-host disease [GVHD], relapse, death)

SECONDARY OUTCOMES:
Time to neutrophil recovery
Primary graft failure
Overall survival
Quality of life
Time to acute GVHD
Time to chronic GVHD
Chronic GVHD details
Cost
Detailed donor and patient self-reported outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Couban, MD, Study Chair — Cancer Care Nova Scotia; Jeffrey H. Lipton, MD, PhD — Princess Margaret Hospital, Canada
Locations (16):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States
- Australia (2):
  - Institute of Medical and Veterinary Science, Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
- Canada (11):
  - Vancouver Hospital and Health Science Center, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Cancer Care Nova Scotia, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Hopital de L'Enfant Jesus, Québec, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
- Auckland City Hospital, Auckland, New Zealand
- King Faisal Specialist Hospital and Research Center, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Kariminia A, Ivison S, Ng B, Rozmus J, Sung S, Varshney A, Aljurf M, Lachance S, Walker I, Toze C, Lipton J, Lee SJ, Szer J, Doocey R, Lewis I, Smith C, Chaudhri N, Levings MK, Broady R, Devins G, Szwajcer D, Foley R, Mostafavi S, Pavletic S, Wall DA, Couban S, Panzarella T, Schultz KR. CD56bright natural killer regulatory cells in filgrastim primed donor blood or marrow products regulate chronic graft-versus-host disease: the Canadian Blood and Marrow Transplant Group randomized 0601 study results. Haematologica. 2017 Nov;102(11):1936-1946. doi: 10.3324/haematol.2017.170928. Epub 2017 Sep 21. PMID 28935847